CLINICAL TRIAL: NCT02540356
Title: A Phase 1/2a, Open-Label, Parallel, Two-Arm Dose-Escalation Study to Assess the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of BAX69 in Subjects With Refractory Ovarian Cancer With Malignant Ascites
Brief Title: Phase 1/2a Two-Arm Dose-Escalation Study of BAX69 in Subjects With Malignant Ascites of Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 391402; 2015-003492-29 (EudraCT Number)
Record Dates: First submitted 2015-08-24; First posted 2015-09-03 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Refractory Ovarian Cancer With Recurrent Symptomatic Malignant Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-Route Arm (Experimental): BAX69 administered weekly by intraperitoneal (IP) infusion only
  Interventions: Biological: BAX69 Single-Route Arm
- Double-Route Arm (Experimental): BAX69 administered weekly by intravenous (IV) infusion + intraperitoneal (IP) infusion
  Interventions: Biological: BAX69 Double-Route Arm

INTERVENTIONS:
Biological: BAX69 Single-Route Arm — Intraperitoneal (IP) only
  Other Names: Macrophage Migration Inhibitory Factor Antibody (Anti-MIF); Imalumab
  Arms: Single-Route Arm
Biological: BAX69 Double-Route Arm — Intravenous (IV) infusion + intraperitoneal (IP) infusion
  Other Names: Imalumab; Macrophage Migration Inhibitory Factor Antibody (Anti-MIF)
  Arms: Double-Route Arm

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of BAX69 monotherapy given either as intraperitoneal (IP) infusion (Single-Route Arm); or as IP infusion after intravenous (IV) infusion (IV+IP) (Double-Route Arm), and to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) for each Arm separately, in subjects with refractory ovarian cancer and recurrent malignant ascites. In both Arms, the plasma pharmacokinetics (PK) of BAX69 will be characterized, and pharmacodynamics (PD) markers will be explored in plasma and ascites. Two expansion cohorts will further assess the tolerability of the RP2D and explore clinical signs of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed informed consent
2. Female participants of non-childbearing potential, ≥18 years of age
3. Anticipated life expectancy >3 months at the time of screening
4. Metastatic ovarian epithelial cancer that are platinum-resistant, and has no better option available in the investigator's opinion
5. Recurrent symptomatic malignant ascites having required at least 2 paracenteses within a 45-day interval prior to baseline paracentesis
6. Participants who have an indwelling draining IP catheter (to be drained only under medical supervision)
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2
8. Adequate hematological function, defined as:

   * Platelet count ≥100,000/μL
   * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) <1.5 times the upper limit of normal (ULN)
   * Absolute neutrophil count ≥1,000/μL
   * Hemoglobin ≥9 g/dL, without the need for transfusion in the 2 weeks prior to screening
9. Adequate renal function, defined as serum creatinine ≤2.0 times ULN and creatinine clearance >50 mL/min or estimated glomerular filtration rate (eGFR) >50 mL/min/1.73 m^2
10. Adequate liver function, defined as:

    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN for participants without liver metastases, or ≤5 times ULN in the presence of liver metastases
    * Bilirubin ≤2.0 times ULN, unless participant has known Gilbert's syndrome
11. Adequate venous access
12. Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Known central nervous system metastasis that is unstable within the last 2 months
2. Prior malignancy within the past 3 years, with the exception of curatively treated basal or squamous cell carcinoma of the skin, ductal carcinoma in situ of breast, in situ cervical carcinoma, and superficial bladder cancer
3. Residual AEs >Grade 2 from previous treatment
4. Myocardial infarction within 6 months prior to C1D1 treatment, and/or prior diagnoses of congestive heart failure (New York Heart Association Class III or IV), unstable angina, unstable cardiac arrhythmia requiring medication; and/or the participant is at risk for polymorphic ventricular tachycardia (eg, hypokalemia, family history or long QT syndrome)
5. Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg confirmed upon repeated measures
6. Left ventricular ejection fraction <50% as determined by echocardiogram (ECHO) performed at screening or within 30 days prior to C1D1
7. QT/QTc interval >480 msec, before C1D1 treatment administration, as determined by screening electrocardiogram (ECG)
8. Received anti-tumor therapy (chemotherapy, investigational product, radiotherapy, retinoid therapy, or hormonal therapy) within 2 weeks (less than 14 days) prior to C1D1 with no residual toxicity >Grade 1; antibody therapy, molecular targeted therapy within 5 half-lives prior to C1D1
9. Major surgery within 4 weeks (less than 28 days) prior to C1D1
10. Active joint inflammation or other immune disorder involving joints (osteoarthritis is not exclusionary)
11. Active infection involving IV antibiotics within 2 weeks prior to C1D1
12. Positive serology test for hepatitis B virus (HBV), hepatitis C virus (HCV), or active tuberculosis
13. Positive serology test for human immunodeficiency virus (HIV) type 1 and 2, or known history of other immunodeficiency disease
14. Participant has received a live vaccine within 2 weeks (less than 14 days) prior to C1D1
15. Known hypersensitivity to any component of recombinant protein production by Chinese Hamster Ovary (CHO) cells
16. Any disorder or disease, or clinically significant abnormality on laboratory or other clinical test(s) (eg, blood tests and ECG), that in medical judgment of the investigator may impede the participant's participation in the study, pose increased risk to the participant, and/or confound the results of the study
17. Participant is a family member or employee of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (6):
- United States (6):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Georgia Regents University, Augusta, Georgia
  - Women's Health Specialists, Silver Spring, Maryland
  - Montefiore Medical Center, The Bronx, New York
  - Stephenson Cancer Center at The University of Oklahoma, Oklahoma City, Oklahoma
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the low number of study participants).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants were enrolled for this study and 1 participant was a screen failure. Study was stopped early with only 1 participant having been dosed.
Groups:
- Single-Route Arm: BAX69 administered weekly by intraperitoneal (IP) infusion as 1 of the following predefined dose regimens: 5mg/kg (Cohort S1), 10mg/kg (Cohort S2), 15mg/kg (Cohort S3)
- Double-Route Arm: BAX69 administered weekly by intravenous (IV) infusion + intraperitoneal (IP) infusion as 1 of the following predefined dose regimens: 5mg/kg IV + 5mg/kg IP (Cohort D1), 10mg/kg IV + 5mg/kg IP (Cohort D2), 10mg/kg IV + 10mg/kg IP (Cohort D3)
Period: Overall Study
Arm/Group | Single-Route Arm | Double-Route Arm
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Terminated due to disease progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Route Arm | Double-Route Arm | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of Dose-limiting Toxicity (DLT)
Description: DLT is defined as any drug related treatment-emergent adverse event that occurs during the 28-day period after the first dose of Imalumab and that meets any of these criteria: - Any ≥ grade 3 non-hematologic toxicity assessed by the investigator as related to study drug (except: single lab value out of normal range not necessarily translating or considered a feature of clinical diagnosis requiring an intervention per investigator's interpretation and resolves to ≤ Grade 2 with adequate measure in 7 days; Transient grade 3 elevations of hepatic transaminases in the absence of simultaneous increase in serum bilirubin; Alopecia) - Any toxicity resulted in dose delay for ≥14 days - Any grade 4 hematologic toxicity (except lymphopenia) - Grade 3 febrile neutropenia - Grade 3 thrombocytopenia associated with bleeding - Any life-threatening complication/abnormality not covered in the NCICTCAE v4.03
Time Frame: 4 weeks
Population: Study was terminated early with only one participant dosed. No statistical analysis was performed on this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Primary Outcome: The Ratio of Puncture Free Survival (PuFS) Over Puncture-free Interval at Baseline
Description: PuFS is defined as the time from the last dose of Imalumab to the first therapeutic paracentesis after that, or death, whichever occurs first. Puncture-free interval at baseline is calculated as the time between the last 2 therapeutic paracenteses immediately before the first dose of Imalubmab.
Time Frame: 4 weeks
Population: Study was terminated early with only one participant dosed. No statistical analysis was performed on this outcome measure. Additionally, due to concerns that the participant would be at risk of being re-identified, study results are not posted.
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Ratio of Time to First Paracentesis Post-treatment Over Puncture-free Interval at Baseline
Description: Time to first paracentesis post-treatment is calculated as the time between the last dose of Imalumab to subsequent first therapeutic paracentesis.
Time Frame: 4 weeks
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Ascites Volume Per Unit Time With Treatment
Description: The volume of ascites from the last dose of Imalumab to the first post-treatment paracentesis per unit time will be compared to the volume of the last pre-treatment paracentesis per unit time. At each paracentesis, the volume of fluid that can be removed safely (measured by ultrasound-guided paracentesis) to achieve close to dryness should be withdrawn, measured, and documented.
Time Frame: Up to 4 weeks
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Ascites-related Symptoms
Description: Ascites related symptoms: anorexia, nausea, early satiety, vomiting, abdominal pain, abdominal swelling, dyspnea, fatigue, swollen ankles, heartburn
Time Frame: Baseline, weekly during the treatment period, and every 2 weeks during the safety follow-up period, up to approximately 6 months)
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs) and/or Treatment-emergent Adverse Events (TEAEs), Regardless of Causality or Relationship to Study Drug
Time Frame: Throughout the study period of approximately 22 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 1 | 0
Participants
  SAEs | 0 | 0
  TEAEs related to study drug | 0 | 0
  TEAEs not related to study drug | 1 | 0

7. Secondary Outcome: Occurrence of Binding and/or Neutralizing Anti-imalumab (BAX69) Antibodies Following Treatment With Imalumab (BAX69)
Time Frame: Throughout the study period of approximately 22 months
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Imalumab (BAX69) Plasma Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax)
Time Frame: Predose; and post-dose at 1.5, 4, 8, 24, and 72 hours
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Imalumab (BAX69) Plasma Pharmacokinetic (PK) Parameter: Minimum Observed Concentration (Cmin)
Time Frame: Predose; and post-dose at 1.5, 4, 8, 24, and 72 hours
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Imalumab (BAX69) Plasma Pharmacokinetic (PK) Parameter: Area Under the Concentration vs Time Curve (AUC)
Time Frame: Predose; and post-dose at 1.5, 4, 8, 24, and 72 hours
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Imalumab (BAX69) Plasma Pharmacokinetic (PK) Parameter: Half-life (t1/2)
Time Frame: Predose; and post-dose at 1.5, 4, 8, 24, and 72 hours
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Imalumab (BAX69) Plasma Pharmacokinetic (PK) Parameter: Apparent Systemic Clearance (CL)
Time Frame: Predose; and post-dose at 1.5, 4, 8, 24, and 72 hours
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Imalumab (BAX69) Plasma Pharmacokinetic (PK) Parameter: Volume of Distribution (V)
Time Frame: Predose; and post-dose at 1.5, 4, 8, 24, and 72 hours
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Quality of Life (QoL) Measure - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Questionnaire
Description: QoL will be assessed using EORTC QLQ-C30.
Time Frame: Weekly from the baseline visit to the last week of safety follow-up (8 weeks or longer, if additional treatment will be implemented)
Population: as for outcome 2
Arm/Group | Single-Route Arm | Double-Route Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of Imalumab (BAX69) until study completion/discontinuation or 56 (±2 days) following the last dose of Imalumab.
Groups:
- Overall Trial: Treatment with Imalumab (BAX69) over a 4-week treatment period administered weekly at one of the following dose regimens: BAX69 5mg/kg IP (intraperitoneal) (Cohort S1), 10mg/kg IP (Cohort S2), 15mg/kg IP (Cohort S3), 5mg/kg IV (intravenous) + 5mg/kg IP (intraperitoneal) (Cohort D1), 10mg/kg IV + 5mg/kg IP (Cohort D2), 10mg/kg IV + 10mg/kg IP (Cohort D3)
Arm/Group | Overall Trial
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Trial (N=1)
Abdominal distention (Grade 2) (Gastrointestinal disorders) | 1 (2)
Hypokalemia (Grade 1) (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Grade 1) (Metabolism and nutrition disorders) | 1 (1)
Right knee pain (Grade 1) (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early with only 1 subject having been dosed. Therefore no statistical analysis was performed on the outcome measures. Only descriptive data for one subject are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until completion of the multi-center publication or twelve months following the conclusion of the study at all sites, whichever is first. Baxalta requires a review of results communication at least 90 days prior to submission. Baxalta may request an additional delay up to 60 days (e.g. for intellectual property protection).